CLINICAL TRIAL: NCT01609894
Title: Individualized Fortification of Breast Milk With Fat, Carbohydrate and Protein for Preterm Infants
Brief Title: Individualized Fortification of Breast Milk
Acronym: IFO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster Children's Hospital (Other)
Responsible Party: Principal Investigator, Christoph Fusch, Professor and Division Head, McMaster Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201205IFO
Record Dates: First submitted 2012-05-30; First posted 2012-06-01 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Postnatal Growth Disorder; Neurodevelopment
Keywords: Postnatal development; Breast milk fortification; Composition of breast milk

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Individualized fortification of breast milk (Experimental): 1. Macronutrient content (for protein, carbohydrate and fat content) will be analyzed of native breast milk batches which had been prepared for 24 hr feeding.
  2. Routine fortifier will be added to breast milk batches.
  3. Modular products for individual adjustment of protein and/or carbohydrate and/or fat will be given in order to achieve target macronutrient level.
  Interventions: Dietary Supplement: Individualized fortification of breast milk
- Routine fortification of breast milk (Active Comparator): 1. Macronutrient content (for protein, carbohydrate and fat content) will be analyzed of native breast milk batches which had been prepared for 24 hr feeding.
  2. Routine fortifier will be added to breast milk batches.
  Interventions: Dietary Supplement: Routine fortification of breast milk

INTERVENTIONS:
Dietary Supplement: Individualized fortification of breast milk — Lactose, fat and protein content will be measured prior to breast milk fortification.
  Subsequently, breast milk for preterm infants will individually fortified adjusted by using data from milk analysis.
  Arms: Individualized fortification of breast milk
Dietary Supplement: Routine fortification of breast milk — Infants will be fed routine fortified breast milk.
  Arms: Routine fortification of breast milk

SUMMARY:
The proposed research will investigate individualized fortification of breast milk based on daily milk analysis of carbohydrate, protein, and fat content in a randomized double blind controlled trial. The combination of additional fat, carbohydrate and protein and commercial fortifier will be added to ensure that the milk contains the target amounts of nutrient. Growth and development of these infants will be compared with that of infants fed mother's milk that has been supplemented with the current standard amounts. The postnatal growth of the infants will be assessed by measuring weight, length and head circumference and fat and lean mass using highly accurate, non-invasive methods throughout the intervention period and at the first follow-up visit after discharge at 3 months. Neurological development will be analyzed at the age of 18 months.

The investigators hypothesize that individualized fortification of breast milk improves the nutritional intake of preterm infants, optimizing growth, and thus this will positively impact neurodevelopment and health.

ELIGIBILITY:
Inclusion criteria:

1. Gestational age < 32weeks (maternal dates or early fetal ultrasound);
2. Tolerating an enteral intake of ≥ 100 ml/kg/d for ≥ 24h;
3. Subject is anticipated to receive the intervention for ≥ 3 consecutive weeks after full enteral feeding (≥ 150 mL/kg/d) has been achieved; and
4. Written informed consent has been obtained from the infant's legal representative.

Exclusion criteria:

1. Infants with intrauterine growth restriction, small for gestational age defined by a weight less than 3rd percentile using sex specific reference data for birth weight
2. Gastrointestinal malformation, major congenital anomalies and chromosomal abnormalities;
3. Babies with enterostoma or short gut syndrome;
4. Necrotizing enterocolitis, defined by feeding intolerance associated with positive x-ray findings (pneumatosis intestinalis - Bell Stage 2; air in the biliary tract or free air in the peritoneum - Bell Stage 3);
5. Renal disease, defined by symptoms (oliguria, anuria, proteinuria, hematuria) associated with an increased blood urea nitrogen 10 mmol/L79 and creatinine of 130 mmol/L80;
6. Hepatic dysfunction, defined by jaundice (direct bilirubin >1.0 mg/dl) that is associated with one or more abnormal liver function tests (AST, ALT or GGT);
7. Participation in another clinical trial that may affect outcomes of this study; or
8. Probability of transfer to another NICU or level II nursery outside the McMaster Children's Hospital before the minimum period of three weeks is completed.

Post-randomisation exclusion criteria:

1. Infants fed more than 25% of mean caloric intake for a consecutive week with formula milk;
2. Fluid restriction < 140mL/kg/d for ≥ 3 consecutive days;
3. Sepsis - all infants with gram-negative sepsis will be removed from the study.

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112 (Estimated)
Dates: Start 2013-08; Primary Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
growth during first three weeks of intervention | first three weeks during intervention before 36 weeks of gestation
  change in body weight gain will be accessed daily.

SECONDARY OUTCOMES:
enteral energy intake | from inclusion at postmentrual age <32 weeks until 36 weeks
  fat, carbohydrate, protein, and caloric intake by enteral feeding will be assesed daily
neurodevelopment | at 18 month corrected age
  Bayley Scales of Infant Development III
weight gain | from inclusion at postmentrual age <32 weeks until 18 month corrected age
  change in body weight [g]
body length | from inclusion at postmentrual age <32 weeks until 18 month corrected age
  change in body length [cm]
head circumference | from inclusion at postmentrual age <32 weeks until 18 month corrected age
  change in head circumference [cm]
body composition | from inclusion at postmentrual age <32 weeks until 3 month corrected age
  change in body composition measured with air displacement plethysmography (body weight, body volume, calculated fat and lean mass)
body composition (bio-electrical impedance analysis) | from inclusion at postmentrual age <32 weeks until 18 month corrected age
  change in body composition measured with bio-electrical impedance analysis (impedance at 5, 50, 100 and 200 kHz, resistance at 50 kHz, reactance at 50 kHz, phase angle at 50 kHz)
skin fold thickness | from inclusion at postmentrual age <32 weeks until 18 month corrected age
  change in skin fold thickness [cm]
feeding intolerance | during intervention (postmentrual age <32 weeks until 36 weeks)
  occurence of feeding intolerance defined by vomitting, bloody gastric residuals, or abnormal abdomen (tender, discolored, absent bowel sounds)
morbidity | during intervention (postmentrual age <32 weeks until 36 weeks)
nutrient's blood parameter | during intervention (postmentrual age <32 weeks until 36 weeks)
  triglycerides, glucose, blood urea nitrogen, blood gases, electrolytes, pH
breast milk analysis | during intervention (postmentrual age <32 weeks until 36 weeks)
  using near-infrared analysis breast milk's macronutrients (fat, lactose and protein) will be measured daily

CONTACTS AND LOCATIONS:
Overall Officials: Christph Fusch, MD, PhD, FRCPC, Principal Investigator — McMaster Children's Hospital
Locations (1):
- Faculty of Health Science, McMaster Children's Hospital, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Fabrizio V, Trzaski JM, Brownell EA, Esposito P, Lainwala S, Lussier MM, Hagadorn JI. Individualized versus standard diet fortification for growth and development in preterm infants receiving human milk. Cochrane Database Syst Rev. 2020 Nov 23;11(11):CD013465. doi: 10.1002/14651858.CD013465.pub2. PMID 33226632
- [Derived] Rochow N, Fusch G, Ali A, Bhatia A, So HY, Iskander R, Chessell L, El Helou S, Fusch C. Individualized target fortification of breast milk with protein, carbohydrates, and fat for preterm infants: A double-blind randomized controlled trial. Clin Nutr. 2021 Jan;40(1):54-63. doi: 10.1016/j.clnu.2020.04.031. Epub 2020 May 6. PMID 32446787